CLINICAL TRIAL: NCT07110649
Title: Experimental Study on the Improvement of Shoulder Range of Motion in College Women Basketball Players by Virtual Reality Technology
Brief Title: Virtual Reality Rehabilitation for Shoulder Injuries in Female College Basketball Players
Acronym: VRSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiarong Wang (Other)
Responsible Party: Principal Investigator, Jiarong Wang, Researcher, Jiarong Wang
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SMAPVC16042024; No External Funding (Other: Sanming Medical and Polytechnic Vocational College)
Record Dates: First submitted 2025-07-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Virtual Reality Therapy
Keywords: VR; shoulder; female basketball player

STUDY DESIGN:
Intervention Model Description: Virtual Reality Rehabilitation Group: Participants in this group will receive immersive virtual reality rehabilitation training aimed at improving shoulder joint mobility and basketball-specific movements.
  Traditional Rehabilitation Group: Participants in this group will undergo conventional physical therapy and manual training for shoulder joint rehabilitation.
  Control Group: Participants in this group will not receive any intervention and will be monitored for natural progression.
  Each group will consist of 15 participants, and the study will last for a total of 9 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Rehabilitation Group (Experimental): Participants in this group will receive immersive virtual reality rehabilitation training, which includes exercises designed to improve shoulder joint range of motion and simulate basketball-specific movements.
  Interventions: Device: Virtual Reality Rehabilitation Group
- Traditional Rehabilitation Group (Active Comparator): Participants in this group will undergo conventional rehabilitation therapy, including manual therapy and exercises aimed at improving shoulder joint mobility.
  Interventions: Other: Traditional Rehabilitation Group
- Control Group (No Intervention): Participants in this group will not receive any rehabilitation intervention and will only be monitored for natural recovery.

INTERVENTIONS:
Device: Virtual Reality Rehabilitation Group — Conducted in three progressive stages using VR games: improving ROM, strengthening shoulder muscles, and simulating game scenarios.
  Other Names: PICO3
  Arms: Virtual Reality Rehabilitation Group
Other: Traditional Rehabilitation Group — Used conventional physical therapy methods based on established rehabilitation programs.
  Arms: Traditional Rehabilitation Group

SUMMARY:
This study aims to evaluate the effectiveness of virtual reality technology in the rehabilitation of shoulder injuries in college women's basketball players. We hypothesise that rehabilitation training using a virtual reality system can improve the range of motion of the shoulder joint more effectively than traditional physical therapy methods and help athletes return to optimal condition. The study will compare the effects of virtual reality training, traditional rehabilitation training, and no intervention group.

DETAILED DESCRIPTION:
To explore the intervention effects of virtual reality (VR) technology in shoulder injuryrehabilitation and its feasibility and practical value in college students 'sports recovery, thisstudy focuses on the theme of "The Therapeutic Effects of Virtual Reality Technology onShoulder lnjuries in Chinese University Basketball Players." A nine-week sports rehabilitationexperimental study was conducted. in line with the policy spirit of integrated development ofphysical education and health in Fujian Province's universities and the research direction ofour university's sports discipline, the project team collaborated with experts both inside andoutside the campus to conduct rehabilitation training experiments for a group of eligible female basketball players from Chinese universities.The study involved 45 female basketball players from universities in Fujian Province, allof whom experienced varying degrees of shoulder joint mobility limitations. Based on theiathletic abilities and injury severity, the participants were randomly divided into three groupsthe VR rehabilitation group, the traditional rehabilitation group, and the control group, with 15participants in each group. The VR rehabilitation group underwent immersive virtual realitytraining, which included exercises to increase joint range of motion and simulate specificbasketball movements. The traditional rehabilitation group received conventional physicatherapy and manual training. The control group did not receive any form of intervention.Statistical methods were used to compare and analyze the effectiveness of differentintervention methods in improving shoulder joint mobility. The experiment also combined on-site rehabilitation records and performance feedback to comprehensively evaluate theapplication prospects of virtual reality rehabilitation in sports medicine.

ELIGIBILITY:
Eligible participants are female college basketball players between the ages of 18 and 24 who have limited shoulder range of motion (ROM limitation) as confirmed by standardized clinical assessment. Participants must regularly engage in basketball training and have no history of shoulder surgery. Individuals will be excluded if they have neurological disorders or other medical conditions that may interfere with virtual rehabilitation, a history of vertigo or intolerance to virtual reality environments, or severe shoulder instability or injuries that prevent participation in rehabilitation training.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Shoulder Joint Range of Motion After 9-Week Rehabilitation | From baseline assessment to the end of 9-week rehabilitation period
  The primary outcome of this study is the change in shoulder joint range of motion (ROM) across five directions: flexion, abduction, extension, internal rotation, and external rotation. Shoulder ROM will be measured using a digital goniometer with ±1° accuracy, following standardised protocols from the American Academy of Orthopaedic Surgeons (AAOS). The normal ROM values for shoulder movement are as follows: Flexion (0°-180°), Abduction (0°-180°), Extension (0°-60°), Internal Rotation (0°-70°), and External Rotation (0°-90°). A positive change indicates an improvement in shoulder joint mobility from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: JIARONG WANG, PHD, Principal Investigator — JIARONGW
Locations (1):
- Sanming Medicaand Polytechnic Vocational College, Sanming, Fujian, China

IPD SHARING:
Plan to Share IPD: No
Due to privacy concerns and the nature of the data, individual participant data will not be shared with other researchers. All data will be kept confidential and used only for the purpose of this study. However, if necessary, data can be made available upon request for academic or research purposes, but will not be shared for commercial use.

REFERENCES:
- [Background] Morikawa LH, Tummala SV, Brinkman JC, Crijns TJ, Lai CH, Chhabra A. Shoulder and Elbow Injuries in National Basketball Association Athletes and Their Effects on Player Performance. Orthop J Sports Med. 2023 Oct 6;11(10):23259671231202973. doi: 10.1177/23259671231202973. eCollection 2023 Oct. PMID 37810744
- See also: Covers standardsStudy Protocol 1. Background and Objective Shoulder injuries are common among athletes, particularly female collegiate basketball players, for various types of disability assessment, especially in the fields of medicine and rehabilitation — https://translate.google.com/
- Available data/document: Individual Participant Data Set: VR_Shoulder_Rehab_2024 — https://translate.google.com/ — This dataset includes the shoulder range of motion (ROM) and visual analogue scale (VAS) pain scores for 45 collegiate female basketball players. The data were collected over a 9-week period as part of a randomized controlled trial evaluating the effectiveness of virtual reality-assisted rehabilitation for shoulder injuries. The dataset is anonymized and can be shared upon request for non-commercial academic research purposes only
- Available data/document: Study Protocol: VR_Shoulder_Rehab_2024 — https://translate.google.com/ — This study aims to evaluate the effect of virtual reality (VR)-assisted rehabilitation training on shoulder range of motion (ROM) and pain relief in college women's basketball players. Forty-five college women's basketball players with shoulder injuries were randomly divided into three groups: VR-assisted rehabilitation group, traditional rehabilitation group, and control group. The VR group underwent 9 weeks of immersive training, the traditional group received conventional physical therapy, and the control group did not receive any intervention. The primary evaluation index was shoulder ROM (flexion, abduction, internal rotation, and external rotation), and the secondary evaluation index was pain intensity (VAS). All assessments will be performed at baseline and after the intervention, and the data will be analyzed using SPSS statistical software. The study hypothesized that VR rehabilitation methods can improve shoulder range of motion, reduce pain, and increase athlete participatio
- Available data/document: Statistical Analysis Plan: VR_Shoulder_Rehab_2024 — https://translate.google.com/ — This study used a randomized controlled method and all randomly assigned participants were included. Data analysis was performed using SPSS or R software. Baseline characteristics will be described using descriptive statistics, with continuous variables expressed as mean ± standard deviation (SD) and categorical variables expressed as frequency/percentage. The primary outcome was shoulder range of motion (ROM), and the difference before and after the intervention was compared using paired t-test (if the data did not conform to normal distribution). The differences between the groups were analyzed using MANOVA, and if the data did not conform to normal distribution, the Kruskal-Wallis test was used. The secondary outcome was pain intensity (VAS), and independent sample t-test or Mann-Whitney U test was used to compare continuous data. Missing data were handled using multiple imputation. The statistical significance level was set at p < 0.05, and 95% confidence intervals and effect sizes
- Available data/document: Informed Consent Form: VR_Shoulder_Rehab_2024 — https://translate.google.com/ — To explore the effect of virtual reality technology on improving the range of motion of the shoulder joints of Chinese college women's basketball players and provide a basis for future sports rehabilitation training. The study has been approved by the Ethics Committee of Sanming Medical Science and Technology Vocational College. Participants will receive 9 weeks of shoulder rehabilitation training, including traditional rehabilitation or virtual reality intervention. During the study, we will collect data on the participants' shoulder range of motion (ROM) and pain scores (VAS), which will only be used for statistical analysis of this study. All personal information and data will be strictly confidential, limited to research purposes, and will not be used for other purposes. Participation in this study is completely voluntary, and participants can withdraw without reason at any stage, and withdrawal will not be affected or punished in any way.
- Available data/document: Data Monitoring Committee Charter: SMMAPVC16042024 — https://translate.google.com/ — This dataset includes data from a 9-week study on VR-assisted rehabilitation for shoulder mobility in female basketball players. The study was approved by the Ethics Review Committee of Sanming Medical and Polytechnic Vocational College (SMMAPVC), with written informed consent obtained from all participants. Data is available for academic research purposes only.
- Available data/document: Clinical Study Report: VR_Shoulder_Rehab_2024 — https://translate.google.com/ — The VR group showed an increase in ROM in flexion from 157.24° to 171.64°, abduction from 157.93° to 173.21°, internal rotation from 57.94° to 67.43°, and external rotation from 71.17° to 84.16° (p < 0.001). The pain score in the VR group also decreased significantly, with the VAS score for flexion decreasing from 6.2 to 3.5, abduction from 6.0 to 3.3, and internal rotation from 5.8 to 3.9 (p < 0.001). In contrast, the traditional rehabilitation group showed some improvement, but the effect was smaller than that of the VR group, and no significant change was observed in the control group. Statistical analysis showed that VR-assisted rehabilitation was superior to traditional methods in improving the range of motion of the shoulder joint and reducing pain, and showed higher rehabilitation participation and motivation. Therefore, VR technology has great application potential in sports rehabilitation for shoulder injuries.

DOCUMENTS (2):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT07110649/Prot_000.pdf
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT07110649/ICF_001.pdf